CLINICAL TRIAL: NCT02649491
Title: Using an Electronic Nose to Predict Gastrointestinal Consequences of Pelvic Radiotherapy
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: University of Warwick (Other)
Responsible Party: Sponsor
Other Study IDs: 4201
Record Dates: First submitted 2015-09-08; First posted 2016-01-07 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Toxicity; Malignancy
Keywords: Radiotherapy; Chemotherapy; Metabonomics; Electronic Sensing; GI Toxicity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will be asked to provide stool and urine samples and complete symptom assessment questionnaires at 6 time points: baseline (before treatment), 2 and 6 weeks after starting radiotherapy, 6 months after completion of radiotherapy and 12 and 24 months after completion of treatment. In addition, patients will be asked to provide a rectal swab and a saliva sample, which will be stored and potentially used at a later stage to characterize any differences in the microbial populations present. (Funding will be sought elsewhere to analyse these samples).
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cohort Observation — Study participation will be offered to women, newly diagnosed with a gynecological malignancy who are due to be treated with pelvic radiotherapy.

SUMMARY:
Scientists have developed an instrument which works like an "electronic nose". It is able to "sniff" smells and separate different smells by their electronic "signature". Studies using an electronic nose strongly suggest that smelling samples taken from humans (e.g. urine/ stool/ sweat/ tears) can identify different electronic smell signature from people with different diseases and in the future might be a new and easier way to diagnose serious conditions at an earlier stage.

In a very small study, it has been successfully shown that using an electronic nose to sniff a stool sample does seem to identify people before they have had any radiotherapy - who will go on to get serious bowel side effects of radiotherapy. If this finding is correct, this is very important as it would allow the cancer doctors the option to change the way they give radiotherapy if they knew that a person was at very high risk of serious side effects from the treatment and to start treatment for the side effects at a much earlier stage.

In this study the investigators want to confirm in a larger study whether the previous findings are correct, and to see whether similar results can be obtained by sniffing urine rather than stool (that would be much easier for everyone) and identify exactly which part of the complicated "smell" signature is different in the people who will get side effects. This may lead for the investigators to able to identify why people are making this specific smell and then do something about changing the smell before treatment starts. The likeliest cause for the production of a smell which predisposes to side effects is a specific group of germs living in the bowel. If these germs can be identified, then there are many possible ways of changing these germ populations in advance of radiotherapy.

Enormous improvements have been made in treating cancer in recent years leading to hugely improved survival, however, treatment not infrequently can lead to side effects. Of all the possible long term physical side effects of cancer treatment, gastrointestinal (GI) symptoms are the most common and can have a great impact on daily activity. It is becoming increasingly clear that development of side effects in the bowel is not just related to the dose and way the radiotherapy is delivered.

DETAILED DESCRIPTION:
There have been enormous improvements in outcomes for patients diagnosed with cancer in recent years. Patients survive longer and the number of survivors after cancer therapy increases 3% annually in the UK and 11% in the USA.It is estimated that there will be 4 million cancer survivors in the UK by 2030.Patients after cancer treatments have many unmet needs which are often caused by the very therapies given to cure or control the cancer. Of all the possible chronic physical side effects of cancer treatment, gastrointestinal (GI) symptoms are the most common and not only have the greatest impact on daily activity but also frequently carry serious financial, psychological and social implications.

During treatment for the cancer, GI symptoms are common and their causes are poorly researched despite their impact on patients' quality of life and the fact that when they occur they often require dose reduction or cessation of chemotherapy and/or radiotherapy with potential impact on outcome. In addition, the GI side effect may not settle once anti-cancer treatment is stopped. In patients receiving radiotherapy for a tumor in the pelvis, more severe acute reactions predispose to worse long term side effects.

At least 17,000 British patients are treated annually with radiotherapy for pelvic cancer. Up to 80% of these patients are left with chronic alteration in GI function, 50% state that this affects their daily activity and 30% that this change in function has a moderate or severe effect. While progress has been made in defining optimal management of chronic changes in bowel function after cancer treatment and UK multi-professional guidance to aid clinicians has been published it would be extremely valuable to be able to predict those in advance who might go on to develop serious problems as a result of radiotherapy so as to have the opportunity to provide them with pre-treatment counseling, potentially modify the cancer treatment and introduce toxicity modifying therapies at the earliest opportunity.

It is widely believed that technical advances in the delivery of radiotherapy will abolish GI problems however, recent compelling data demonstrate that 30% of patients treated with "perfect" radiotherapy - meeting every described constraint still develop significant un-predicted problems. While mechanisms by which gastrointestinal symptoms occur after cancer treatment are starting to be understood and personal parameters which change the risk profile for individuals are being identified (body mass index, concomitant chemotherapy, use of a statin or ACE inhibitor, the presence of diabetes mellitus, hypertension, connective tissue disorders or HIV infection) the reasons why some patients remain symptom free whilst others experience severe side effects remains under researched.

It has become clear that development of GI toxicity is not solely related to the dose and way the radiotherapy is delivered, and a phenomenon independent of the radiation called the 'the consequential effect' is a second reason why some people get chronic side effects after radiotherapy. An important driver of the 'consequential effect' is increasingly believed to be the microbiota, the vast numbers of bacteria that live in our guts. The gastrointestinal microbiota are a complex ecosystem of up to 1,000 bacterial species in any one individual. The species vary greatly between individuals but within each individual, the flora composition remains stable for the majority of the species over time. The diversity of the microbiota is high in healthy people and low in people with GI side effects after pelvic radiotherapy, a process which very closely parallels findings in people with other much more intensively researched inflammatory conditions of the bowel.

Normal gut flora produce gases from their metabolites (Volatile Organic Compounds or VOCs). The gold standard for analyzing volatile organic compounds is gas chromatography/mass spectrometry (GCMS).

GCMS analyses gasses to identify all chemical components of that gas. However, this is very expensive and requires a specialized laboratory to process the samples hence is not a viable option in day to day clinical practice.

Two alternative techniques can be applied to analyse those VOCs: electronic sensing (e-nose) or High Field Asymmetric Ion Mobility Spectrometry (FAIMS).

Electronic sensing techniques are applied via an instrument (electronic nose) that attempts to replicate the biological olfactory system, by investigating samples as a whole, instead of identifying specific chemicals within a complex sample. The air above the sample (head space) is drawn into the e-nose and passed across an array of chemical sensors. The size of the array varies, but most are between 6 and 32 sensors. As each sensor is dissimilar, the interaction between the sensor and the sample is unique and an olfactory signature for this complex odor can be created.

Fields Asymmetric Waveform Ion Mobility Spectometry (FAIMS) is a new technology capable of separating gas phase ions at atmospheric pressure and at room temperature. As with the electronic nose, FAIMS can be used for the real time analysis of complex chemical components, looking at the total chemical composition of a sample. Differences in the way the ionised molecules move in high electric fields are used to draw a mobility signature of a complex sample.

The e-nose and FAIMS techniques have been used successfully in small studies to diagnose lung disease, diabetes, bladder cancer, tuberculosis, cyanide poisoning, renal failure and schizophrenia. Focusing on gastrointestinal disorders, consistent changes in the VOCs produced by patients with inflammatory bowel disease, bile acid malabsorption, gastrointestinal cancer, coeliac disease, Clostridium difficile infection can be identified compared to healthy individuals.

In a paper published in 2012 of a retrospective blinded pilot study using the e-nose in 23 patients in whom the investigators analysed stool samples collected immediately before the start of radiotherapy. Of the 23 patients selected, 11 subsequently had minimal or no side effects from radiotherapy and 12 had severe toxicity. The e-nose analysed the samples and astonishingly identified with 100% accuracy two completely distinct groups of patients: those who would develop severe toxicity during radiotherapy and those who would not. The results of this study suggest that the substantial differences in the volatile gases produced by stool samples in the two populations, have a critical impact on toxicity and the reason that different fermentation products occur is either because the microbiological composition of stool differs between the two groups, or because bacterial function is somehow different. Whatever the reason, these findings suggests that the microbiota plays a critical role in the initiation of radiation induced inflammation are completely consistent with findings from other studies using very complex methodologies and with studies investigating the role of the microbiota in other GI conditions .

ELIGIBILITY:
Inclusion Criteria

* Patients aged 18 years or above able to give informed consent
* Patients to be treated with radical, adjuvant or neo-adjuvant radiotherapy for a new diagnosis of a gynaecological cancer.
* Ability of the patient to provide informed consent.

Exclusion Criteria

* Patients aged less than 18 years
* Patients who are pregnant
* Patients unable to give informed consent
* Patients being treated privately
* Patients due to have their post-treatment follow-up elsewhere in the country
* Patients on studies with conflicting end-points

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 2 years we will recruit 120 patients undergoing radical radiotherapy for a new, histologically proven, gynaecological malignancy at the Royal Marsden Hospital. Patients will be followed up for 2 years after completion of radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in Olfactory Signatures in patient sample | 24 months
  A 6 point difference in the olfactory signatures in different samples (rectal swab, stool sample,urine, sample saliva sample) between patients who develop severe toxicity* and those with no or minimal toxicity.

SECONDARY OUTCOMES:
Changes in Bristol Stool Chart Parameters. | 24 months
  The Bristol stool chart categorizes the types of stool a person passes into 7 categories. It is a helpful tool to assess stool consistency in combination with other tools assessing GI symptoms, however it does not describe the severity of toxicity so no cut off values.
Changes in the scores of Inflammatory Bowel Questionnaire, | 24 months
  For IBDQ a higher score will indicate a better Quality of Life (QoL). A change in IBDQ will indicate the level of patients QoL over the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jervoise Dr Andreyev, MA, Phd, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom